CLINICAL TRIAL: NCT06360198
Title: The Relationship Between Posture, Sense of Position, Musculoskeletal Discomfort and Anxiety in Asymptomatic Individuals: A Cross-Sectional Study
Brief Title: The Relationship Between Posture, Sense of Position, Musculoskeletal Discomfort and Anxiety
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-874/08
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Kyphosis Postural Thoracic; Proprioception; Musculoskeletal System; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: The only group of this cross-sectional observational study consists of individuals over the age of 18. There were no orthopedic and neurological chronic diseases included. Individuals with severe visual and hearing problems and individuals who had undergone surgery within the last 6 months were excluded.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was applied to the group.

SUMMARY:
It is known that posture is affected by various factors such as somatosensation, visual perception and cognition. In addition, it is also thought to affect conditions such as stress and anxiety through receptors. The aim of this study was to investigate the relationship between postural changes such as thoracic kyphosis, musculoskeletal problems, trunk position sense and anxiety in young individuals who were asymptomatic in terms of musculoskeletal problems.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Volunteered to participate in the study
* No systemic or neurological disease

Exclusion Criteria:

* Severe visual and hearing problems
* Orthopedic injury or surgery in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young people who are asymptomatic in terms of musculoskeletal problems
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Throcic Kyphosis | Baseline
  The thoracic kyphosis angle was evaluated with a dual digital inclinometer (Acumar, Lafeyette, USA). Repetitive cervical flexion, extension and lateral flexion movements were asked from the subjects before the measurement. They were also asked to perform back rotation of the shoulders and to take a deep breath in and out. Subsequently, they were asked to stand in a normal position in which they were comfortable and the measurement was performed. The inclinometer was placed on the T1-2 and T12-L1 vertebrae. The value on the inclinometer screen was noted as the degree of kyphosis. A kyphosis angle of 20-40 degrees is considered normal. Values above 45 degrees are considered as hyperkyphosis.

SECONDARY OUTCOMES:
Trunk Position Sense | Baseline
  Trunk position sense was evaluated with a dual digital inclinometer (Acumar, Lafeyette, USA) during 30 degrees of trunk flexion. For the measurement, the subjects were asked to stand in a standing and comfortable position. The inclinometer was placed on the T1 and S1 vertebrae. Individuals were asked to perform 30 degrees of trunk flexion with their eyes closed. The measurement was taught by performing 2 trials. Then, the individuals were asked to find the target angle that was taught. The angle that the individuals thought was the target angle was recorded. The difference between the recorded angle and the target angle was written as absolute value. The process was repeated three times and averaged. There is no specific reference value for trunk flexion position sensation.
Musculoskeletal Discomfort | Baseline
  Musculoskeletal disorders of the individuals were assessed with the Cornell Musculoskeletal Disorder Scale. The scale consists of three categories assessing the frequency, severity and work intervention of musculoskeletal discomfort in 20 different body parts within a week. The answers given in the frequency section are scored between 0-1.5-3.5-5-10. In the severity of musculoskeletal discomfort and the work disability caused by the musculoskeletal system disorder sections the answers are scored between 1-3. The scores for each body part are multiplied and then summed to obtain a total score from the three sections. The total score is the sum of all section scores. A lower score indicates less musculoskeletal discomfort.
Anxiety | Baseline
  Anxiety of the individuals was assessed with the Generalised Anxiety Disorder-7 scale. The scale evaluates the experiences in the last 2 weeks. The Generalised Anxiety Disorder-7 scale is a four-point Likert-type scale based on self-report. The total score is obtained by adding the score of the answer given to each item. The higher the total score obtained from the scale, the higher the level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No